CLINICAL TRIAL: NCT05327192
Title: Collection of Samples From Women Diagnosed With Vulvovaginal Candidiasis for Validation of Vaginal Microbiome Analysis Method
Brief Title: VVC Sampling Study for Analysis Validation
Status: Completed | Type: Observational
Sponsor: Gedea Biotech AB (Industry)
Responsible Party: Sponsor
Other Study IDs: CL4-2
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Vulvovaginal Candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Vaginal samples to study bacterial DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention, only sampling — No intervention

SUMMARY:
This is a biomarker multi-centre study to validate an extraction method of fungal and bacterial DNA extracted from vaginal swabs from adult women with confirmed VVC.

The study population will consist of post-menarchal, pre-menopausal females, 18 years or older, seeking care for VVC symptoms.

Vaginal samples will be examined under a microscope for yeast forms (hyphae or pseudohyphae) or budding yeast. If the Investigator assesses that the patient has VVC, based on examination and the potassium hydroxide (KOH) test, two vaginal secretion samples will be collected by a vaginal swab. One sample will be cultured to verify the presence of Candida and the other will be used for sequencing analysis of the vaginal microbiome.

Samples from a total of 10 women are planned to be taken.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women aged 18 years or older
2. Diagnosis of VVC, defined as having a white or creamy vaginal discharge plus the following findings:

   1. At least 2 of the following signs and symptoms of VVC that are characterized as at least moderate: itching, burning, irritation, edema, redness, or excoriation.
   2. Potassium hydroxide (KOH) or saline preparation from the inflamed vaginal mucosa or secretions revealing yeast forms (hyphae or pseudohyphae) or budding yeasts.
3. Having decisional capacity and providing written informed consent
4. Signed informed consent and willing and able to comply with all study requirements

Exclusion Criteria:

None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of post-menarchal, pre-menopausal females, 18 years or older, seeking care for VVC symptoms.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
Correlation between vaginal sample DNA sequencing and VVC confirmed by clinical diagnosis and culture. | 1 day

OTHER OUTCOMES:
Evaluate resolution of bacterial DNA sequencing using 16S regions. | 1 day

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Research and Development Department, Berkshire Healthcare NHS Foundation Trust, Slough

IPD SHARING:
Plan to Share IPD: No